CLINICAL TRIAL: NCT06431217
Title: Investigating for Immunological Correlates of Protection Against Invasive Group B Streptococcus Disease in Infants Less Than 90 Days of Age.
Brief Title: Group B Strep Correlates of Protection Study
Acronym: GBSCoP
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: University of KwaZulu (Other); University of Stellenbosch (Other); University of Pretoria (Other); University of Cape Town (Other)
Responsible Party: Principal Investigator, Farzanah Laher, Doctor, University of Witwatersrand, South Africa
Other Study IDs: GBS CoP
Record Dates: First submitted 2019-03-05; First posted 2024-05-28 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Maternal Health; Child Health; Infectious Diseases
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood, Vaginal Swab collection, cord blood collection, DBS collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Streptococcus agalactiae or Group B Streptococcus (GBS) is a leading cause of neonatal sepsis in developed and developing countries.

The study aims to bolster the evidence base of establishing a sero-correlate of protection against invasive GBS disease in infants.

These sero-correlates of protection will be used to study the effectiveness of GBS vaccine against invasive disease.

DETAILED DESCRIPTION:
Observational Case-Control Study

* A cohort of 15,000 mother-infant dyads will be enrolled at Chris Hani Baragwanath Academic Hospital (n=10,000) and Rahima Moosa Mother and Child Hospital(n=5,000) over an 18-24-month period, anticipated to start in the first quarter of 2019.
* Enrolment into the cohort study will occur at antenatal clinic, during the early stages either of labour or immediately post-delivery.
* In parallel, enrolment of GBS cases will occur at the time of diagnosis of invasive GBS disease. These "retrospective cases" will be enrolled at multiple facilities across South Africa.
* Infants will be followed up until 89 days of age to identify cases of suspected sepsis and hospitalizations.

Determine the infant GBS serotype Ia and III specific capsular serum IgG antibody level associated with 80% reduced odds of invasive GBS disease between 0-89 days of age for the combined "cohort" and "retrospectively enrolled" cases.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women attending for antenatal care at one of the participating antenatal-clinics and/or delivering at CHBAH or RMMCH.
2. Subjects aged ≥18 years.
3. Able to understand and comply with planned study procedures.
4. Provides written informed consent.

Exclusion Criteria:

1. Refusal to consent to study participation.
2. Receipt of any blood products in the past 4 weeks or anticipated during labour.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 5.1.1. Cohort population Maternal-newborn dyads enrolled at CHBAH or RMMCH prior to or during delivery-admission, from whom maternal and cord blood are collected.
  5.1.2. Control population Controls will be defined as newborns born to mothers enrolled into the cohort study, whose mother is colonized by a serotype homologous to that of a case to which they matched, but who do not develop invasive GBS disease within 90 days of life. Cases and controls will matched by serotype, gestational age (34-<37 weeks and ≥37 weeks gestation) and maternal age (<25 years, 25-<35 years and ≥35 years). Maternal HIV infection status will be assessed as an effect modifier.
Sampling Method: Non-Probability Sample
Enrollment: 17842 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Primary Objective | 1 - 1.5 years
  Determine the infant GBS serotype Ia and III specific capsular serum IgG antibody level associated with 80% reduced odds of invasive GBS disease between 0-89 days of age for the combined "cohort" and "retrospectively enrolled" cases. Anti-CPS IgG concentrations were determined with the use of a quantitative direct immunoassay (Luminex) that measured levels of antibodies binding to CPS serotypes Ia, Ib, and II through V.

CONTACTS AND LOCATIONS:
Locations (1):
- Rmpru/Vpd, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No